CLINICAL TRIAL: NCT06373081
Title: A Clinical Study on the Safety and Efficacy of Anti-CD19-CD3E-CAR-T Cells in the Treatment of Relapsed or Refractory Autoimmune Disease
Brief Title: Anti-CD19-CD3E-CAR-T Cells in Relapsed/Refractory Autoimmune Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Changzheng Hospital (Other)
Responsible Party: Principal Investigator, Xu huji, Professor and Chief Physician, Head of the Department of Rheumatology and Immunology, Shanghai Changzheng Hospital., Shanghai Changzheng Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CD19-CD3E-CN-A1
Record Dates: First submitted 2024-04-15; First posted 2024-04-18 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Systemic Lupus Erythematosus (SLE); Sjogren's Syndrome; Systemic Sclerosis; Inflammatory Myopathy; ANCA Associated Vasculitis; Antiphospholipid Syndrome
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Sjogren's Syndrome; Scleroderma, Systemic; Myositis; Anti-Neutrophil Cytoplasmic Antibody-Associated Vasculitis; Antiphospholipid Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Anti-CD19-CD3E-CAR-T Cells treatment (Experimental): Anti-CD19-CD3E-CAR-T cells, Autologous T-cells expressing a chimeric antigen receptor directed to CD19.
  Interventions: Biological: Anti-CD19-CD3E-CAR-T cells

INTERVENTIONS:
Biological: Anti-CD19-CD3E-CAR-T cells — The injection of anti-CD19-CD3E chimeric antigen receptor T (CAR-T) cells, referred to as anti-CD19-CD3E-CAR-T cells. The anti-CD19-CD3E-CAR protein is composed of a murine-derived CD19 single-chain variable fragment (scFv) FMC63, CD28 hinge and transmembrane regions, the intracellular domain of CD3E, the intracellular domain of CD28, and the intracellular domain of CD3ζ, all linked in sequence.

SUMMARY:
This is an investigator-initiated trial to evaluate the safety and efficacy of anti-CD19-CD3E-CAR-T cells in the relapse or refractory autoimmune diseases.

DETAILED DESCRIPTION:
This is an investigator-initiated trial to evaluate the safety and efficacy of anti-CD19-CD3E-CAR-T cells in the relapse or refractory autoimmune diseases.

Study intervention consists of a single infusion of CAR-transduced autologous T cells administered intravenously after a lymphodepleting therapy regimen consisting of fludarabine and cyclophosphamide.

Interim analysis will be performed when participants finish the visit of 12 weeks after CAR-T cells infusion.

ELIGIBILITY:
Step 1. Assessment of eligibility for Enrollment Inclusion Criteria for Enrollment

Common Inclusion Criteria:

1. Age between 18 and 65 years old (inclusive), regardless of gender.
2. Positive expression of CD19 on peripheral blood B cells confirmed by flow cytometry.
3. Functional requirements for major organs are as follows: 1) Bone marrow function must meet: A. Neutrophil count ≥ 1×109/L (no colony-stimulating factor treatment within 2 weeks before examination); B. Hemoglobin ≥ 60g/L; 2) Liver function: Alanine aminotransferase (ALT) ≤ 3×ULN (excluding ALT elevation due to inflammatory myopathy), aspartate aminotransferase (AST)≤3×Upper limit of normal (ULN) (excluding AST elevation due to inflammatory myopathy), TBIL≤1.5×ULN (or ≤ 3.0×ULN for subjects with Gilbert syndrome); 3) Renal function: creatinine clearance rate (CrCl) ≥ 30ml/minute (calculated by Cockcroft/Gault formula, acute CrCl decrease due to the target disease is excluded); 4) Coagulation function: International standardized ratio (INR) <1.5×ULN, prothrombin time (PT) <1.5×ULN; 5) Cardiac function: Stable hemodynamic.
4. Female subjects of childbearing potential and male subjects with partners of childbearing potential must use medically approved contraception or abstinence during the study treatment period and for at least 6 months after the end of the study treatment; Female subjects of childbearing potential must have a negative Human chorionic gonadotropin (HCG) test within 7 days before study enrollment and not be lactating.
5. Willing to participate in this clinical study, sign an informed consent form, have good compliance, and cooperate with follow-up.

Disease-Specific Inclusion Criteria

Refractory/Relapsed SLE:

1. SLE fulfilling the 2019 the American College of Rheumatology (ACR) /European League Against Rheumatism (EULAR) and classification criteria.
2. Systemic lupus erythematosus disease activity index (SLEDAI)-2000 score ≥ 6 with at least one BILAG (British Isle Lupus Rating Group Index 2004) A or two BILAG B; or SLEDAI-2000 score ≥ 8.
3. Definition of relapsed/refractory: Conventional treatment over 6 months remains ineffective, or disease recurrence after remission. Definition of conventional treatment: the use of glucocorticoids and cyclophosphamide, and any one or more of the following immunomodulatory drugs: antimalarials, azathioprine, mycophenolate mofetil, methotrexate, leflunomide, tacrolimus, cyclosporine, and biologics including belimumab, rituximab, and tocilizumab, etc.

Refractory/Relapsed Sjogren's syndrome:

1. Primary Sjogren's syndrome fulfilling the 2002 AECG criteria or the 2016 ACR/EULAR classification criteria.
2. EULAR Sjögren's Syndrome Disease Activity Index (ESSDAI) ≥ 6
3. Positive anti-SSA/Ro antibodies
4. Definition of relapsed/refractory: Conventional treatment over 6 months remains ineffective, or disease recurrence after remission. Definition of conventional treatment: the use of glucocorticoids and cyclophosphamide, and any one or more of the following immunomodulatory drugs: antimalarials, azathioprine, mycophenolate mofetil, methotrexate, leflunomide, tacrolimus, cyclosporine, and biologics including belimumab, rituximab, and tocilizumab, etc.

Refractory/Relapsed/Progressive Systemic Sclerosis:

1. Scleroderma fulfilling the 2013 ACR classification criteria
2. Positive scleroderma-related antibodies.
3. Presence of diffuse cutaneous sclerosis or active interstitial lung disease (high-resolution computed tomography (HRCT) showing ground-glass opacities);
4. Definition of relapsed/refractory: Conventional treatment over 6 months remains ineffective, or disease recurrence after remission. Definition of conventional treatment: the use of glucocorticoids and cyclophosphamide, and any one or more of the following immunomodulatory drugs: antimalarials, azathioprine, mycophenolate mofetil, methotrexate, leflunomide, tacrolimus, cyclosporine, and biologics including belimumab, rituximab, and tocilizumab, etc.
5. Definition of progressive: Rapid skin progression (mRSS increase > 25%); or progression of lung disease (forced vital capacity (FVC) decrease by 10%, or FVC decrease by more than 5% with diffusing capacity of the lung for carbon monoxide (DLCO) decrease by 15%).

Note: Meeting either criterion 4 or 5 is sufficient.

Refractory/Relapsed/Progressive Inflammatory Myopathy:

1. Inflammatory myopathy fulfilling the 2017 EULAR/ACR classification criteria (including Dermatomyositis (DM), Polymyositis (PM), Anti-Synthetase Syndrome (ASS), and Necrotizing Myopathy (NM)).
2. Positive myositis antibodies;
3. Muscle involvement with Manual Muscle Testing-8 (MMT-8) score less than 142 and at least two abnormalities found among the following five core measurements (Physician Global Assessment (PhGA), Patient Global Assessment (PtGA), or extramuscular disease activity score ≥ 2; Health Assessment Questionnaire (HAQ) total score ≥ 0.25; muscle enzyme levels ≥ 1.5×ULN; or MMT-8 ≥ 142, but with active interstitial lung disease (HRCT showing ground-glass opacities);
4. Definition of relapsed/refractory: Conventional treatment over 6 months remains ineffective, or disease recurrence after remission. Definition of conventional treatment: the use of glucocorticoids and cyclophosphamide, and any one or more of the following immunomodulatory drugs: antimalarials, azathioprine, mycophenolate mofetil, methotrexate, leflunomide, tacrolimus, cyclosporine, and biologics including belimumab, rituximab, and tocilizumab, etc.
5. Definition of progressive: Rapid progression of interstitial lung disease within a short period.

Note: Meeting either criterion 4 or 5 is sufficient.

Refractory/Relapsed ANCA-Associated Vasculitis:

1. ANCA-Associated Vasculitis fulfilling 2022 ACR/EULAR criteria, including microscopic polyangiitis, granulomatosis with polyangiitis, and eosinophilic granulomatosis with polyangiitis.
2. Positive ANCA-associated antibodies (MPO-ANCA or PR3-ANCA positive).
3. The Birmingham Vasculitis Activity Scale (BVAS) ≥ 15 points (a total score of 63 points), indicating active vasculitis.
4. Definition of refractory/relapsed: Conventional treatment over 6 months remains ineffective, or disease recurrence after remission., or disease recurrence after remission. Definition of conventional treatment: the use of glucocorticoids and cyclophosphamide, and any one or more of the following immunomodulatory drugs: antimalarials, azathioprine, mycophenolate mofetil, methotrexate, leflunomide, tacrolimus, cyclosporine, and biologics including belimumab, rituximab, and tocilizumab, etc.

Refractory/Relapsed/Catastrophic Antiphospholipid Syndrome:

1. Primary antiphospholipid syndrome fulfilling 2006 Sydney criteria.
2. Positive phospholipid antibodies with medium to high titers (IgG/IgM for Lupus Anticoagulant (LA), Beta-2 Glycoprotein 1 (B2GP1), or Anticardiolipin (aCL), positive more than twice within 12 weeks).
3. Definition of refractory/relapsed: Standard treatment with warfarin anticoagulation or alternative vitamin K antagonist therapy (maintaining treatment-required INR) or standard therapeutic dose of low molecular weight heparin (LMWH) and use of steroids and cyclophosphamide for recurrent thrombosis;
4. Catastrophic antiphospholipid syndrome needs to meet the following four criteria: (1) involvement of three or more organs, systems, and/or tissues; (2) symptoms occurring within one week; (3) histological confirmation of small vessel occlusion in at least one organ or tissue; (4) positive aPL antibodies.

Note: Meeting either criterion 3 or 4 is sufficient.

Exclusion Criteria:

1. Subjects with a history of severe drug allergies or allergic tendencies;
2. Presence or suspicion of uncontrolled or treatment-required fungal, bacterial, viral, or other infections;
3. Subjects with central nervous system diseases caused by autoimmune diseases or non-autoimmune diseases (including epilepsy, psychosis, organic brain syndrome, cerebral vascular accidents, encephalitis, central nervous system vasculitis);
4. Subjects with insufficient cardiac function;
5. Subjects with congenital immunoglobulin deficiencies;
6. History of malignancy within five years;
7. Subjects with end-stage renal failure;
8. Subjects who are positive for hepatitis B surface antigen (HBsAg) or hepatitis B core antibody (HBcAb) with peripheral blood HBV DNA >ULN; subjects positive for hepatitis C virus (HCV) antibody and peripheral blood HCV RNA; individuals positive for human immunodeficiency virus (HIV) antibody; individuals positive for syphilis testing;
9. Subjects with psychiatric disorders and severe cognitive impairments;
10. Subjects who have participated in other clinical trials within the past 3 months prior to enrollment;
11. Subjects who have received biologics with therapeutic effects for indications within 4 weeks prior to enrollment;
12. Subjects who have received immunosuppressive agents with therapeutic effects for indications within 2 weeks prior to enrollment;
13. Subjects who have received >10mg/d prednisone or equivalent dose of other steroids within 2 weeks prior to enrollment;
14. Pregnant women or women planning to conceive;
15. Subjects whom the investigator believes have other reasons that make them unsuitable for inclusion in this study.

Step 2. Assessment of eligibility for CAR-T Cells Infusion Inclusion Criteria

1. Completion of Step 1 and successful preparation of CAR-T cell product;
2. Adequate organ function, defined as: 1) Creatinine clearance rate (Cockcroft and Gault) >30 mL/min/1.73 m2, excluding acute decrease in CrCl due to the target disease; 2) ALT/AST ≤ 3×ULN (excluding liver enzyme elevation caused by inflammatory diseases); TBIL ≤ 1.5×ULN (Gilbert's syndrome allows TBIL ≤ 3×ULN).

Exclusion Criteria

1. Systemic fungal, bacterial, viral, or other infection that is not controlled (defined as exhibiting ongoing signs/symptoms related to the infection and without improvement, despite appropriate antibiotics or other treatment);
2. >10mg/d prednisone or equivalent dose of other steroids within 72 hours prior to CAR-T infusion.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2024-04-20 (Estimated); Primary Completion 2025-04-15 (Estimated); Study Completion 2026-04-15 (Estimated)

PRIMARY OUTCOMES:
The incidence of dose-limiting toxicities (DLTs) (Safety) | Up to 28 days from CAR-T infusion
  Safety assessments, including the incidence of dose-limiting toxicities (DLTs) in patients receiving CAR-T cells, are conducted using the NCI-CTCAE version 5.0 standards.
Proportion of patients for whom the desired dose of anti-CD19-CD3E-CAR-T cells can be successfully manufactured | Up to 21 days from apheresis
  Proportion of patients for whom the desired dose of anti-CD19-CD3E-CAR-T cells can be successfully manufactured
Clinical response for relapsed/Refractory SLE | 12 weeks post CAR-T infusion
  SLE Response Index 4 (SRI-4) response: Min/Max Value: Not specified; a decrease in score indicates improvement; higher scores indicate worse outcome.
Clinical response for Sjögren's Syndrome | 12 weeks post CAR-T infusion
  Sjögren's tool for assessing response (STAR): Min/Max Value: Not specified; a decrease in score indicates improvement; higher scores indicate worse outcome.
Clinical response for relapsed/refractory/progressive systemic sclerosis | 12 weeks post CAR-T infusion
  Composite Response Index in Systemic Sclerosis (CRISS): Min/Max Value: 0 to 1 (expressed as a probability); closer to 1 indicates a better response; higher scores indicate better outcome.
Clinical response for relapsed/refractory/progressive inflammatory myopathy | 12 weeks post CAR-T infusion
  Total Improvement Score (TIS):Min/Max Value: Not specified; an increase in score indicates improvement; higher scores indicate better outcome.
Clinical response for relapsed/refractory anti-neutrophil cytoplasmic antibody (ANCA)-associated vasculitis: | 12 weeks post CAR-T infusion
  Birmingham vasculitis activity score (BVAS) score:Min/Max Value: 0 to 63; an increase in score indicates worsening condition; higher Scores Indicate: Worse Outcome.
Clinical response for relapsed/refractory/Catastrophic Antiphospholipid Syndrome | 12 weeks post CAR-T infusion
  Evaluation of new thrombosis as an indicator of relapsed/refractory/catastrophic Antiphospholipid Syndrome; higher scores Indicate worse outcome (indicates progression of the syndrome).

CONTACTS AND LOCATIONS:
Overall Officials: Huji Xu, Ph.D, MD, Principal Investigator — Shanghai Changzheng Hospital
Locations (1):
- Shanghai ChangZheng hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No
Due to concerns regarding the security of patient personal information.